CLINICAL TRIAL: NCT04941313
Title: A Single-blind, Randomized, and Placebo-Controlled Phase 1 Study to Evaluate the Safety and Tolerability of 3D-229 by Intravenous Single Dose Escalation and Repeated Doses in Healthy Subjects
Brief Title: Phase 1 Study of 3D229 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 3D Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3D229-CN-001
Record Dates: First submitted 2021-05-31; First posted 2021-06-28 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-03

CONDITIONS: Healthy Subject

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single Dose Escalation-3D229 (Experimental): two sequential dose escalation cohorts - patients are randomized either to investigational drug or matching placebo
  Interventions: Drug: 3D229
- Single Dose Escalation- placebo (Placebo Comparator): two sequential dose escalation cohorts - patients are randomized either to investigational drug or matching placebo
  Interventions: Other: Placebo
- Repeat Dose-3D229 (Experimental): Four single doses of the investigational drug or matching placebo - patients are randomized either to investigational drug or matching placebo
  Interventions: Drug: 3D229
- Repeat Dose-placebo (Placebo Comparator): Four single doses of the investigational drug or matching placebo - patients are randomized either to investigational drug or matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 3D229 — 3D229 is an investigational drug.
  Arms: Repeat Dose-3D229; Single Dose Escalation-3D229
Other: Placebo — Matching placebo
  Arms: Repeat Dose-placebo; Single Dose Escalation- placebo

SUMMARY:
This is a Phase 1 Study to Evaluate the Safety and tolerability of 3D-229 in health subjects

DETAILED DESCRIPTION:
A Single-blind, Randomized, and Placebo-Controlled Phase 1 Study to Evaluate the Safety and tolerability of 3D-229 by Intravenous Single Dose Escalation(SAD) and Repeated Doses(RD) in Healthy Subjects. A SAD portion of the study consists of 2 sequential dose escalation cohorts, whereas RD portion of the study consists of a single cohort receiving 4 weekly doses of 3D229. In both SAD and RD study arms, subjects are randomized to receive either a study intervention (3D229) or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects had no clinically significant condition or disease confirmed by medical history, medical assessment, physical examination, clinical laboratory tests, and 12-lead electrocardiogram (ECG) at screening and on the day prior to the first study drug administration;
2. Male or female, aged 18-55 years at the time of signing the informed consent form;
3. Body mass index (BMI) between 18 and 30 kg/m 2 (Containing 18 and 30 kg/m 2 ) within range;
4. Negative urine drug screen/alcohol breath test at screening and 1 day prior to first study drug administration;
5. Has not used tobacco products (including nicotine patches/gum) within 3 months prior to screening and agrees to avoid such products throughout the study;
6. Complete abstinence for at least 14 days prior to the first dose of study drug and Take effective contraceptive measures within 3 months after the last dose(including Complete abstinence、 barrier contraception and completed sterilization operation), no fertility, sperm donation, egg donation program
7. If the subject is female, the serum pregnancy test at screening and urine pregnancy test on the day before first dose should be negative;
8. Ability to fully read, understand and sign the informed consent form;
9. Ability to communicate adequately with the investigator and to comply with the requirements of the entire study.

Exclusion Criteria:

1. Blood pressure ≥ 140/90 mmHg or pulse > 100 beats/min at rest at screening;
2. QT interval corrected for heart rate using Fridericia ' s formula (QTcF) > 430 msec (males) and > 450 msec (females) at screening;
3. Pregnant or lactating women;
4. Males with partners in pregnancy;
5. Concurrently enrolled in another clinical trial, or received any study drug within 3 months prior to the first dose (or 5 drug half-lives, whichever is longer);
6. Subject has a history of drug or alcohol abuse or dependence within the past 1 year;
7. Use of any prescription or over-the-counter medications, including analgesics, hormonal contraceptives (oral contraceptives or implanted contraceptives), natural food supplements, or dietary/herbal supplements (including vitamins), 14 days or 5 drug half-lives, whichever is longer;
8. Donation of more than 200 mL of blood within 56 days prior to the first dose, or planned to donate blood during the study until 1 month after completion of the study;
9. Hepatitis B virus (HBV) surface antigen, hepatitis C virus antibody (HCV), or human immunodeficiency virus (HIV) test results are currently or ever positive;
10. Prior or current condition that, in the opinion of the investigator, may affect the conduct of the study or observations (to be confirmed by medical history);
11. History or current patient ' s clinically significant disease,Including but not limited to: active tuberculosis, asthma, angioedema, bronchospasm, ulcerative disease, gastrointestinal hemorrhage, coagulation disorder, hypertension, edema, heart failure, hypokalemia, hyperkalemia, cardiovascular disease, hypersensitivity to any biological agent, and significant impact on immune responseSevere skin diseases or other conditions of the force;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of 3D229-Adverse events | Up to 7 weeks
  Monitoring of adverse events

SECONDARY OUTCOMES:
AUC | Up to 7 weeks
  Area under the curve
Cmax | Up to 7 weeks
  Maximum observed concentration
Ctrough | Up to 7 weeks
  Serum concentration observed at end of a single dose and observed pre-dose during repeat doses
Tmax | Up to 7 weeks
  Time to reach maximum observed plasma concentration
λz | Up to 7 weeks
  Terminal phase elimination rate constant
t1/2 | Up to 3 weeks
  Terminal half-life
CL | Up to 7 weeks
  The total body clearance
V | Up to 7 weeks
  Volume of distribution
serum GAS6 | Up to 7 weeks
  evaluate the serum GAS6 level

CONTACTS AND LOCATIONS:
Overall Officials: xueying ding, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General hospital, Shanghai, Hongkou District, China

IPD SHARING:
Plan to Share IPD: No